CLINICAL TRIAL: NCT04580446
Title: HYHOPE: Phase I Study of De-intensified Hypofractionated Radiation Therapy for Human Papilloma Virus-associated Oropharynx Cancer
Brief Title: HYHOPE: De-intensified Hypofractionated Radiation Therapy for HPV-associated Oropharynx Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Principal Investigator, Dominic Moon, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-1079
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Human Papillomavirus-Related Carcinoma; Oropharyngeal Cancer
Keywords: Radiation Dose Hypofractionation
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Rolling 6 dose finding cohort followed by dose expansion cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated radiotherapy with concurrent chemotherapy (weekly cisplatin 40 mg/m2) (Experimental): Level 0: 46.5 Gy in 15 fractions, 5 fractions/week
  Level -1: 52 Gy in 20 fractions, 5 fractions/week
  Interventions: Radiation: Hypofractionated intensity modulated radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated intensity modulated radiotherapy — Hypofractionated intensity modulated radiotherapy with concurrent chemotherapy (weekly cisplatin)

SUMMARY:
This is a single arm Phase I study of de-intensified hypofractionated radiation therapy for favorable human papilloma virus-associated oropharynx cancer. It will evaluate the tolerability of a de-intensified hypofractionated radiation therapy regimen completed in 3 weeks (with equivalent biologically effective dose to 60 Gy in 30 fractions) with concurrent weekly cisplatin.

DETAILED DESCRIPTION:
Standard of care radiation therapy (RT) for head and neck squamous cell carcinoma (HNSCC) involves conventional fractionation delivered over a course of 7 weeks. Although hypofractionated RT (HFRT) delivering higher dose of RT each day over a shorter overall treatment time has been studied and adopted as standard of care in many disease sites including breast and prostate cancers, data on HFRT in HNSCC is limited.

There is a strong radiobiological rationale for HFRT for HNSCC to decrease the overall treatment time and thus the effects of accelerated repopulation in this disease entity. In addition, if similar outcomes can be achieved with a reduced number of fractions, cost effectiveness of care can be improved while minimizing the disruption to the patient's personal and professional lives. A substantial decrease in treatment time may improve compliance and financial toxicity associated with the patient's oncologic treatment.

The global COVID-19 pandemic is highlighting the health risk to society at large of having no viable alternative to a 7 week daily RT course for HNSCC, especially in the setting of compromised immune systems associated with concurrent chemotherapy frequently used in this patient population. Thus, the study of HFRT for HNSCC is both timely and potentially paradigm changing for practices across the United States.

The incidence of human papilloma virus (HPV)-associated oropharynx cancer is increasing in the United States, now accounting for 70-80% of all oropharynx cancers. It has a favorable prognosis vs. non-HPV-associated cancers and studies are ongoing to determine the best strategy to de-intensified therapy while maintaining good oncologic outcomes.

The purpose of this single-arm Phase I study is to assess the tolerability and signal for efficacy of de-intensified HFRT for favorable HPV-associated oropharynx cancer. De-intensification will be achieved in two ways. First, the equivalent biologically effective dose (BED) of HFRT used on trial will be 60 Gy of conventionally fractionationated RT (vs. the current standard of care of 70 Gy). Second, the elective nodal volume irradiated will be limited to involved nodal levels and one immediately adjacent level (vs. the current standard of care of entire bilateral neck nodal regions). Patients will complete RT in 15 fractions (3 weeks) with concurrent weekly cisplatin on dose level 0. If a 3-week regimen is not well-tolerated, a 20 fraction regimen will be used on dose level -1.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically-proven diagnosis of T1-3 (up to 6 cm), N0-2 (AJCC 8th edition) p16 positive squamous cell carcinoma of the oropharynx (except T1-2N0 as noted in the exclusion criteria)
2. ≤10 pack-year smoking history and not actively smoking
3. Age ≥18 years
4. ECOG performance status 0-2 or Karnofsky Performance Status 50-100
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
6. Negative serum or urine pregnancy test within 2 weeks before registration for women of childbearing potential.
7. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Distant metastasis
2. T1-2N0 (AJCC 8th edition) p16 positive squamous cell carcinoma of the oropharynx (candidates for definitive RT alone or surgery alone)
3. Inability to receive concurrent weekly cisplatin due to comorbid conditions
4. Synchronous non-skin cancer primaries outside of the oropharynx, oral cavity, larynx, and hypopharynx except for low- and intermediate-risk prostate cancer and well-differentiated thyroid cancer. For prostate cancer, patient should not be receiving active treatment. For thyroid cancer, thyroid surgery may occur before or after radiation treatment, provided all other eligibility criteria are met.
5. Prior invasive malignancy with an expected disease-free interval of less than 3 years
6. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation fields
7. Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the chemotherapy agents in this study
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
10. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
11. History of severe immunosuppression, including HIV, organ or autologous or allogeneic stem cell transplant, or active immunosuppressive medication at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose escalation phase: hypofractionated radiotherapy with cisplatin: Level 0: 46.5 Gy in 15 fractions, 5 fractions/week
  Hypofractionated intensity modulated radiotherapy with concurrent chemotherapy (weekly cisplatin)
- Dose expansion phase: hypofractionated radiotherapy with cisplatin: 46.5 Gy in 15 fractions, 5 fractions/week
  Hypofractionated intensity modulated radiotherapy with concurrent chemotherapy (weekly cisplatin)
Period: Overall Study
Arm/Group | Dose escalation phase: hypofractionated radiotherapy with cisplatin | Dose expansion phase: hypofractionated radiotherapy with cisplatin
Started | 6 | 18
Completed | 6 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation Phase: Hypofractionated Radiotherapy With Cisplatin; Dose Expansion Phase: Hypofractionated Radiotherapy With Cisplatin: 46.5 Gy in 15 fractions, 5 fractions/week, with (weekly cisplatin 40 mg/m2)
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase: Hypofractionated Radiotherapy With Cisplatin | Dose Expansion Phase: Hypofractionated Radiotherapy With Cisplatin | Total
Number analyzed (Participants) | 6 | 18 | 24
Age, Customized [Mean (Full Range); unit: years]
  Age (median range) | 59.6 [52 to 72] | 58.9 [50 to 77] | 59.5 [52 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 18 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: White | 4 | 14 | 18
  Race/ethnicity: Hispanic | 1 | 0 | 1
  Race/ethnicity: African American | 1 | 0 | 1
  Race/ethnicity: Asian | 0 | 1 | 1
  Race/ethnicity: Other/unknown | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 18 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose/Fractionation of Hypofractionated Radiation Therapy
Description: The number of participants experiencing dose-limiting toxicities (DLTs) will be used to determine the maximally tolerated dose (MTD) or optimal fractionation of hypofractionated radiation therapy.
  Level 0: 46.5 Gy in 15 fractions Level -1: 52 Gy in 20 fractions
Time Frame: 3 months
Population: Patients were enrolled using a rolling 6 design at dose level 0 (46.5 Gy in 15 fractions). Enrollment was paused to assess dose-limiting toxicity (DLT; grade 4 toxicity or persistent grade 3 mucositis ≤ 3 months post-treatment). Dose level 0 was evaluated for DLT occurrence. Following this, an expansion cohort was opened, bringing total enrollment to 24 participants. No participants were enrolled at dose level -1 (52 Gy in 20 fractions).
Measure: Count of Participants; unit: Participants
Groups:
- Hypofractionated radiotherapy with concurrent chemotherapy: Level 0: 46.5 Gy in 15 fractions, 5 fractions/week
  Hypofractionated intensity modulated radiotherapy with concurrent weekly cisplatin 40 mg/m2
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
Number analyzed (Participants) | 6
Participants | 0
Statistical Analysis 1: Comparison: Hypofractionated radiotherapy with concurrent chemotherapy; Estimation Parameter: Maximally Tolerated Dose/Fractionation Description: The maximally tolerated dose (MTD)/fractionation of hypofractionated radiation therapy was determined based on the incidence of dose-limiting toxicities (DLTs) observed during the dose-escalation phase. Estimate: 46.5 Gy × 15 fractions; Test type: Other — Descriptive analysis used to identify the dose level associated with ≤1 of 6 participants experiencing a dose-limiting toxicity (DLT), consistent with standard 3+3 design methodology; Maximally Tolerated Dose/Fractionation = 46.5 — MTD/fractionation determined as 46.5 Gy in 15 fractions based on incidence of DLTs during dose escalation (3 + 3 design)

2. Secondary Outcome: Clinician-reported Acute Toxicities
Description: Toxicities as measured by CTCAE v5.0
Time Frame: 0-3 months
Measure: Number; unit: Participants
Groups:
- Hypofractionated radiotherapy with concurrent chemotherapy (weekly cisplatin 40 mg/m2): 46.5 Gy in 15 fractions, 5 fractions/week
  Dose escalation and dose expansion cohorts combined
  Hypofractionated intensity modulated radiotherapy with concurrent weekly cisplatin 40 mg/m2
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy (weekly cisplatin 40 mg/m2)
Number analyzed (Participants) | 24
Participants
  Odynophagia/sore throat (grade 2) | 18
  Oral mucositis (grade 2) | 15
  Weight loss/anorexia (grade 2) | 13
  Dysphagia ( grade 2) | 11
  Dysgeusia (grade 2) | 9
  Xerostomia (grade 2) | 7
  Nausea/vomiting (grade 2) | 2
  Odynophagia/sore throat (grade 3) | 1
  Oral mucositis (grade 3) | 5
  Weight loss/anorexia (grade 3) | 2
  Dysphagia (grade 3) | 2
  Nausea/vomiting (grade 3) | 1

3. Secondary Outcome: Clinician-reported Late Toxicities
Description: As measured by CTCAE v5.0
Time Frame: 3-12 months
Measure: Number; unit: Participants
Groups:
- Hypofractionated radiotherapy with concurrent chemotherapy: 46.5 Gy in 15 fractions, 5 fractions/week
  Dose escalation and dose expansion cohorts combined
  Hypofractionated intensity modulated radiotherapy with concurrent weekly cisplatin 40 mg/m2
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
Number analyzed (Participants) | 24
Participants
  Dysphagia (grade 2) | 1
  Weight loss/anorexia (grade 2) | 1
  Xerostomia (grade 2) | 1
  Grade 3 AE | 0
  Grade 4 AE | 0
  Grade 5 AE | 0

4. Secondary Outcome: Percentage of Participants With Locoregional Control
Description: Locoregional control defined as freedom from locoregional recurrence. Locoregional recurrence defined as biopsy-proven viable cancer originating from the primary tumor site (i.e. oropharynx) or a lymph node basin above the clavicles.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
Number analyzed (Participants) | 24
percentage of participants | 86.2 [68 to 96.8]

5. Secondary Outcome: Percentage of Participants With Progression Free Survival
Description: Progression-free survival defined as time from start of treatment to time of progression or death.
Time Frame: 1-12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
Number analyzed (Participants) | 24
percentage of participants | 82 [59 to 93]

6. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Overall survival defined as time from start of treatment o time of death.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
Number analyzed (Participants) | 24
percentage of participants | 95.8 [74 to 99]

7. Secondary Outcome: Swallowing-related Patient-reported Quality of Life
Description: Change from baseline in swallowing-related quality of life, as measured by the MD Anderson Dysphagia Inventory (MDADI) total score, assessed at specified time points (baseline,1, 3, 6, and 12 months) during and after treatment. Higher scores indicate better function, 0-100. Analyses were descriptive, and a paired t test was used to compare questionnaire results over time with P < .05 considered statistically signiﬁcant. MDADI composite score difference of 10 was deemed clinically meaningful.
Time Frame: 1-12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
Number analyzed (Participants) | 24
score on a scale
  Baseline | 86.5 (13.7)
  1 mo | 77.9 (11.6)
  3 mo | 85.5 (11.3)
  6 mo | 87.8 (12.3)
  12 mo | 89.4 (9.4)

8. Secondary Outcome: Head and Neck Patient-reported Quality of Life
Description: Change from baseline in head and neck patient-reported outcomes quality of life, as measured by the University of Washington Quality of Life questionnaire (UW-QOL), assessed at specified time points (baseline,1, 3, 6, and 12 months) during and after treatment. Higher scores on UW-QOL subscales indicate better quality of life, 0 being worst and 100 being the best outcome. A paired t test was used to compare questionnaire results over time with P < .05 considered statistically signiﬁcant. UW-QOL was divided into 2 subscales of physical and social-emotional function with change of 0.5 x standard deviation (SD) and 0.8 x SD considered moderate and large effect, respectively.
  Scale title: Patient-reported quality of life at baseline and after treatment (0-100) Physical UW-QOL minimum: 45.83 Physical UW-QOL maximum: 100 Social-Emotional UW-QOL minimum: 17.5 Social-Emotional UW-QOL maximum: 100
Time Frame: 1-12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
Number analyzed (Participants) | 24
score on a scale
  Physical Baseline | 93.4 (9.9)
  Physical 1 mo | 74.9 (11.4)
  Physical 3 mo | 80.3 (11.3)
  Physical 6 mo | 84.8 (11.7)
  Physical 12 mo | 85.3 (11.7)
  Social-Emotional Baseline | 89.4 (16.5)
  Social-Emotional 1 mo | 79.9 (10.3)
  Social-Emotional 3 mo | 87.6 (10.0)
  Social-Emotional 6 mo | 90.0 (13.8)
  Social-Emotional 12 mo | 92.1 (10.4)

9. Secondary Outcome: General Patient-reported Quality of Life
Description: EuroQol-5 dimensions (EQ-5D-5L): 1-5, higher scores mean worse quality of life. Index score: 0-1, higher scores mean better quality of life. Visual Analog scale: 0-100, higher scores mean better quality of life.
Time Frame: 1-12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
Number analyzed (Participants) | 24
score on a scale
  Index score Enrollment | 0.916 (0.163)
  Index score 1 mo | 0.879 (0.107)
  Index score 3 mo | 0.909 (0.120)
  Index score 6 mo | 0.915 (0.166)
  Index score 12 mo | 0.933 (0.103)
  Visual Analog Scale Enrollment | 86.8 (12.4)
  Visual Analog Scale 1 mo | 79.1 (11.5)
  Visual Analog Scale 3 mo | 81.9 (12.0)
  Visual Analog Scale 6 mo | 86.1 (9.8)
  Visual Analog Scale 12 mo | 88.9 (8.0)

10. Secondary Outcome: Feeding Tube Dependence
Description: Dependence on tube feeds defined as any participant with daily use of ≥2 nutritional supplements per day via the feeding tube at the time of evaluation.
Time Frame: 1-12 months
Measure: Number; unit: participants
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
Number analyzed (Participants) | 24
participants
  Acute follow up period | 2
  Late follow up period | 1

ADVERSE EVENTS:
Time Frame: 1 year post radiation treatment.
Description: All-Cause Mortality was assessed for 2 year post radiation treatment. Serious and Other Adverse Events were assessed for 1 year post radiation treatment.
Groups:
- Hypofractionated radiotherapy with concurrent chemotherapy: 46.5 Gy in 15 fractions, 5 fractions/week
  Dose escalation and dose expansion cohorts combined. Both cohorts received 46.5 Gy in 15 fractions so the data are combined.
  Hypofractionated intensity modulated radiotherapy with concurrent weekly cisplatin 40 mg/m2
Arm/Group | Hypofractionated radiotherapy with concurrent chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/24
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hypofractionated radiotherapy with concurrent chemotherapy (N=24)
Thromboembolic event bilateral pulmonary embolism (Vascular disorders) | 1
Death NOS (General disorders) | 1 — Motor vehicle accident
Fever (General disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Dysphagia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hypofractionated radiotherapy with concurrent chemotherapy (N=24)
Abdominal Pain (Gastrointestinal disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Allergic reaction (Immune system disorders) | 4
Allergic rhinitis (Reproductive system and breast disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 8
Amnesia (Nervous system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 17
Anosmia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Atrial fibrillation (Cardiac disorders) | 4
Atrioventricular block first degree (Cardiac disorders) | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Blood and lymphatic system disorders - Other, Lymphoma (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, Easy bruising/bleeding (Blood and lymphatic system disorders) | 1
Blurred vision (Eye disorders) | 1
Bood and lymphatic system disorders-Other, Enlarged lymph nodes (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other, bradycardia (Cardiac disorders) | 1
Cardiac disorders - Other, Coronary artery disease (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Cholesterol high (Investigations) | 1
Congenital, familial and genetic disorders - Other, Pure hypercholesterolemia (Congenital, familial and genetic disorders) | 1
Constipation (Gastrointestinal disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Depression (Psychiatric disorders) | 3
Dermatitis radiation (Injury, poisoning and procedural complications) | 24
Diarrhea (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 7
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 24
dry skin (Skin and subcutaneous tissue disorders) | 1
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 24
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 23
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Ear and labyrinth disorders - Other, Ear discharge (Ear and labyrinth disorders) | 1
Ear and labyrinth disorders - Other, Hearing loss (Ear and labyrinth disorders) | 1
Ear and labyrinth disorders - Other, Total cerumen impaction (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 9
Eczema (Skin and subcutaneous tissue disorders) | 1
Edema limbs (General disorders) | 3
Edema Face (General disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Eye disorders - Other, Discharge (Eye disorders) | 1
Eye infection (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Facial pain (General disorders) | 4
Fatigue (General disorders) | 23
Fever (General disorders) | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flu like symptoms (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8
Gastrointestinal disorders - Other, heart burn (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, sputum production (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, change in bowel movement (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, Globus sensation (Gastrointestinal disorders) | 4
Gastrointestinal disorders - Other, Thick secretions (Gastrointestinal disorders) | 7
Gastrointestinal disorders - Other, Tongue swelling (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, Dry throat (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, Gastric pain (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, peri-rectal abscess (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, Tongue pain (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, Cold sores (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, Increased secretions (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, Odynophagia (Gastrointestinal disorders) | 24
Gastrointestinal disorders - Other, Mucus production (Gastrointestinal disorders) | 2
General disorders and administration site conditions - Other, Dislocated shoulder (General disorders) | 1
General disorders and administration site conditions - Other, Speech change (General disorders) | 2
General disorders and administration site conditions - Other, Cold intolerance (General disorders) | 1
General disorders and administration site conditions - Other, Heat intolerance (General disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Hearing impaired (Ear and labyrinth disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Hyperlipidemia (Metabolism and nutrition disorders) | 8
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 19
Hyperthyroidism (Endocrine disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Infections and infestations - Other, COVID-19 (Infections and infestations) | 6
Infections and infestations - Other, Hepatitis B infection (Infections and infestations) | 1
Injury, poisoning and procedural complications - Other, Oropharyngeal erythema (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, Extravasation injury (Injury, poisoning and procedural complications) | 1
Insomnia (Psychiatric disorders) | 6
Investigations - Other, Hematocrit decreased (Investigations) | 1
Investigations - Other, Red Blood Cell decreased (Investigations) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Lung infection (Infections and infestations) | 2
Lymphedema (Vascular disorders) | 8
Lymphocyte count decreased (Investigations) | 8
Malaise (General disorders) | 1
Metabolism and nutrition disorders - Other, Frequent thirst (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, Appetite change (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, Type II Diabetes Mellitus (Metabolism and nutrition disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 22
Musculoskeletal and connective tissue disorder - Other, Left neck mass (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, Herniated disc (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, Neck stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Myocardial infarction (Cardiac disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Nausea (Gastrointestinal disorders) | 19
Neck edema (General disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 9
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nervous system disorders - Other, Temperature sensitivity (Nervous system disorders) | 1
Nervous system disorders - Other, Neuropathy (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 1
Oral Pain (Gastrointestinal disorders) | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Paresthesia (Nervous system disorders) | 2
Periodontal disease (Gastrointestinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rectal fissure (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other, Nocturia (Renal and urinary disorders) | 2
Reproductive system and breast disorders - Other, Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other, Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, Orthopnea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, Snoring (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory, thoracic and mediastinal disorders - Other, Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Retinal detachment (Eye disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other, Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Erythema (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Diaphoresis (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Hair sensitvity (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, Itchiness (Skin and subcutaneous tissue disorders) | 1
Skin infection (Skin and subcutaneous tissue disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 23
Spasticity (Nervous system disorders) | 1
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 2
Surgical and medical procedures - Other, bilateral inguinal herniainguin (Surgical and medical procedures) | 1
Surgical and medical procedures - Other, Fistulectomy anal (Surgical and medical procedures) | 1
Surgical and medical procedures - Other, Root Canal (Surgical and medical procedures) | 1
Surgical and medical procedures - Other, Feeding tube (Surgical and medical procedures) | 1
Testosterone deficiency (Endocrine disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Thrush (Infections and infestations) | 7
Thyroid stimulating hormone increased (Investigations) | 2
Tinnitus (Ear and labyrinth disorders) | 10
Toothache (Gastrointestinal disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 5
Urinary frequency (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Vascular disorders - Other, Aneurysm (Vascular disorders) | 2
Vascular disorders - Other, Aortic atherosclerosis (Vascular disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Weight gain (Investigations) | 1
Weight loss (Investigations) | 18
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
White blood cell decreased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT04580446/Prot_SAP_000.pdf